CLINICAL TRIAL: NCT03380273
Title: AO Multicenter Intervention Trial to Evaluate the Impact of a Bundle of Measures for the Prevention of Surgical Site Infection in Fracture Patients
Brief Title: AO Multicenter Intervention Trial for Prevention of Surgical Site Infection
Acronym: AOPOSSI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment too small and slow due to pandemic situation
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AOPOSSI
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: During two years, patients with fractures are recorded and the occurence of surgical site infections (SSI) in these patients is monitored in different sites over the world. After two years, a bundle of known prevention measures are teached and enforced in these sites. Then the occurence of SSI in fracture patients is monitored for another two years to see whether the bundle decreased the SSI occurence.
Masking Description: It is that preventino measures are enforced in the hospital. This will apply to all patients and no masking is required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-intervention (No Intervention): The number of SSI are collected in this phase. Patients with fractures are enrolled and their standard of care treatment is observed.
- post-intervention (Other): Here the same observations are made as in the first arm, however this is after the hospital staff was thought the prevention measures (all by themselves approved) and enforced to be applied.
  Interventions: Behavioral: Implementation of the AO Trauma SSI Prevention Bundle

INTERVENTIONS:
Behavioral: Implementation of the AO Trauma SSI Prevention Bundle — AOT SSI Prevention Bundle
  Preventive measure
  1. Antibiotic prophylaxis
  2. Perioperative antibiotics
  3. Oxygen administration
  4. Patient temperature
  5. Surgeon protective wear
  6. Patient operative skin preparation
  7. Suction drains
  8. Blood glucose level
  9. Red cell transfusion
  10. Dressing changes
  Arms: post-intervention

SUMMARY:
This study is designed to collect data from 8,476 fracture patients during a pre-and post-intervention phases of two years length each. The intervention consists on the implementation of the AOT SSI Prevention Bundle.

D

DETAILED DESCRIPTION:
During the first phase of the study, 4,238 patients will be recruited and the baseline incidence of surgical site infection at each participating site will be determined. At the beginning of the third year, the bundle will be implemented and data on 4,238 additional patients will be collected. The incidence rate on surgical site infection before and after the intervention will be compared. We hypothesize that this intervention will reduce the infection rate within the first 3 months after surgery from 6% to 4.5% (5% to 3.75% in closed fractures and from 10% to 7.5% in open fractures).

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years

  * Recent fracture (< 10 days) located in femur, tibia or humerus

    * Any type of open or closed fracture
    * Produced by high or low energy trauma
  * Primary fracture treatment with surgery and use of any of the following:

    * Intramedullary or extramedullary devices including cases in which a temporary external fixator is used
    * Joint replacement
  * Informed consent obtained (if required by local EC/IRB), i.e.:

    * Ability to understand the content of the patient information/ICF
    * Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
    * Signed and dated EC/IRB approved written informed consent

Exclusion Criteria:

* Pathologic fracture secondary to tumors, infection or cysts
* Patients with an underlying chronic, bone and joint infection or prior history of a bone and joint infection
* Refracture and non-union
* Peri-implant fractures
* Patients with terminal illness
* Pregnancy or women planning to conceive within the study period
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Infection Rate | within 3 months after surgery
  Surgical site infection rate as defined by CDC or FRI definition

SECONDARY OUTCOMES:
Implementation success of the AOT SSI Prevention Bundle | up to 48 months
  Compliance rate for each measure of the bundle before and after the intervention
Evaluation of attitudes, perception and knowledge concerning SSI | up to 48 months
  Cross sectional survey of surgeons at participating sites performed before and after the implementation of the AOT SSI Prevention Bundle
Surgeon satisfaction | up to 48 months
  Cross sectional survey of opinion concerning user friendliness of the AOT SSI Prevention Bundle, value of the educational intervention and intention to adopt the AOT SSI Prevention Bundle long term before and after its implementation
Health-economic analysis | up to 48 months
  The clinical effectiveness of the implementation of the AOT SSI Prevention Bundle and consecutively the costs saved by preventing infections and its treatment is compared against the costs which have to be invested in order to implement the AOT SSI Prevention Bundle (e.g. costs generated by development of teaching material, time needed to teach/implement the intervention, extra material needed according to the interventions etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kates, MD, Principal Investigator — VCU Health
Locations (14):
- United States (8):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Kentucky Healthcare, Lexington, Kentucky
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Saint Louis University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Germany (2):
  - University Hospital Gießen, Giessen
  - University Hospital Regensburg, Regensburg
- Spitalul Clinic de Urgenta Floreasca, Bucharest, Romania
- Korea University Guro Hospital, Seoul, South Korea
- Hospital Universitari Parc Tauli, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data. The analyses will be done based on groups and these data will be published and shared